CLINICAL TRIAL: NCT01981343
Title: A Randomized, Double Blind, Placebo Controlled Parallel Study Evaluating the Effect of A-F Betafood® on Gallbladder and Liver Function.
Brief Title: A Parallel Study Evaluating the Effect of A-F Betafood® on Gallbladder and Liver Function.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: KGK Science Inc. (Industry)
Collaborators: Standard Process Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 12AGHS
Record Dates: First submitted 2013-11-05; First posted 2013-11-11 (Estimated); Last update posted 2018-04-11 (Actual); Status verified 2018-04

CONDITIONS: Gallbladder
Keywords: Gallbladder motility; A-F Betafood; Betaine; Ejection fraction; Ejection rate; Ultrasound

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- A-F Betafood (Experimental): Two A-F Betafood tablets taken with a meal, 3 times daily for 12 weeks
  Interventions: Dietary Supplement: A-F Betafood
- Placebo (Placebo Comparator): 2 Placebo tablets taken with a meal, 3 times daily for 12 weeks
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: A-F Betafood
  Arms: A-F Betafood
Other: Placebo
  Arms: Placebo

SUMMARY:
Gallstone formation is multifactorial: immutable risk factors include genetics and ethnicity, age and being female, and mutable risk factors include obesity, and metabolic syndrome, diet, rapid weight loss, and other conditions such as cirrhosis, Crohn's disease, irritable bowel syndrome, gallbladder stasis, and the use of certain drugs like Ceftriazone. Previous studies have linked serum cholesterol, and low-density lipoprotein cholesterol levels and fatty liver disease to gallbladder disease. Given betaine's reported beneficial effects on fatty liver and lipid profile, A-F Betafood® may have a beneficial effect on gallbladder function.

The objective of the study is to assess the effect of A-F Betafood® on gallbladder and liver function as measured by gallbladder ultrasounds and liver function tests. The hypothesis is that A-F Betafood® will improve gallbladder and liver function after the 12 week treatment period.

This is a single-center, randomized, double-blind, placebo-controlled, parallel group study with two arms. This study will consist of a single 12 week treatment period. The planned sample size for this study is 50 overweight female subjects, with 25 subjects randomized equally to each of the two study arms in double-blind manner at a ratio of 1:1

ELIGIBILITY:
Inclusion Criteria:

* Females 40-75 years of age or older not of child bearing potential. Defined as females who have had a hysterectomy or oophorectomy, bilateral tubal ligation or are post-menopausal (natural or surgically with > 1 year since last menstruation).OR Female subject of childbearing potential must agree to use a medically approved method of birth control and have a negative urine pregnancy test result
* BMI of 25.0 kg/m2 to 29.9 kg/m2
* Agrees to comply with study procedures
* Healthy as determined by laboratory results, medical history and physical exam
* Has given voluntary, written, informed consent to participate in the study
* Gastrointestinal distress with various fatty foods as determined by the modified GSRS questionnaire
* Family history of gallbladder disease or previous history of gallbladder attacks
* Has a normal resting heart rate 50-80bpm

Exclusion Criteria:

* Women who are pregnant, breastfeeding, or planning to become pregnant during the course of the trial
* Unstable psychiatric disorder requiring hospitalization within past 6 months
* Use of prescription medications, over the counter medications or natural health products/dietary supplements known to affect gastric/gastrointestinal function within 4 weeks of randomization
* Presence of gallstones as determined by ultrasound
* Uncontrolled hypertension defined as untreated systolic blood pressure > 160 mmHg and/or diastolic blood pressure > 100 mmHg
* Clinically significant abnormal laboratory results at screening including: AST, ALT and/or bilirubin > 2 x the ULN; Serum creatinine >1.5 x the ULN or eGFR < 60; Hemoglobin < 123 g/L
* Participation in a clinical research trial within 30 days prior to randomization
* Allergy or sensitivity to test article ingredients, soy, dairy, egg, wheat, peanut, tree nuts, fish or shellfish.
* Individuals who are cognitively impaired and/or who are unable to give informed consent
* Any other condition which in the Investigator's opinion may adversely affect the subject's ability to complete the study or its measures or which may pose significant risk to the subject

Ages: 40 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2013-11-11 (Actual); Primary Completion 2018-02-01 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
Gallbladder and Liver function | 12 weeks
  Changes in Gallbladder Ultrasound and Liver function tests (fasting serum AST, ALT, GGT and hsCRP)

SECONDARY OUTCOMES:
Gastrointestinal distress | 12 weeks
  Modified GSRS questionnaire
Fasting Lipid Profile | 12 weeks
  Changes in serum LDL-C, HDL-C, total cholesterol and triglycerides
Fasting Oxidized LDL | 12 weeks
  Changes in serum oxidized LDL levels
Fasting TNF-alpha | 12 weeks
  Changes in serum TNF-alpha levels
Fasting Adiponectin | 12 weeks
  Changes in serum adiponectin levels
Blood Pressure | Over 12 weeks
  Changes in mean office blood pressure
Heart Rate | Over 12 weeks
  Changes in mean heart rate
Biometrics: weight and BMI | Over 12 weeks
  Changes in mean weight and BMI
Blood Safety Parameters | Over 12 weeks
  Changes in complete blood count, electrolytes (Na, K, Cl), creatinine, eGFR, AST, ALT,GGT, bilirubin
Fasting Malonyldialdehyde | 12 weeks
  Changes in serum malonyldialdehyde (MDA) levels
Adverse events | Over 12 weeks
  Record and monitor any adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Tetyana Pelipyagina, MD, Principal Investigator — KGK Science Inc.
Locations (1):
- KGK Synergize Inc., London, Ontario, Canada